CLINICAL TRIAL: NCT06724614
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Multi-dose Study to Evaluate the Efficacy and Safety of VDPHL01 in Male Subjects With Androgenetic Alopecia
Brief Title: Efficacy and Safety of VDPHL01 in Males With AGA
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Veradermics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 250-13951-302
Record Dates: First submitted 2024-12-04; First posted 2024-12-09 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Androgenetic Alopecia; AGA; Male Pattern Baldness
Keywords: Hair Loss; Male Hair Loss
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- VDHPL01 BID (Experimental): VDPHL01 will be taken orally twice a day, once in the AM and once in the PM.
  Interventions: Drug: VDPHL01
- VDPHL01 QD and Placebo QD (Experimental): Placebo will be taken orally once a day in the AM or PM. VDPHL01 will be taken orally once a day in the AM or PM.
  Interventions: Drug: VDPHL01
- Placebo BID with treatment extension to VDPHL01 BID (Placebo Comparator): Placebo will be taken orally twice a day, once in the AM and once in the PM for the first 6 months of the study. After month 6, VDPHL01 will be taken orally twice a day, once in the AM and once in the PM.
  Interventions: Drug: Placebo
- Placebo BID with treatment extension to VDPHL01 QD and Placebo QD (Placebo Comparator): Placebo will be taken orally twice a day, once in the AM and once in the PM for the first 6 months of the study. After month 6, placebo will be taken orally once a day in the AM or PM. VDPHL01 will be taken orally once a day in the AM or PM.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VDPHL01 — VDPHL01 Extended Release (ER) Tablet
  Arms: VDHPL01 BID; VDPHL01 QD and Placebo QD
Drug: Placebo — Placebo
  Arms: Placebo BID with treatment extension to VDPHL01 BID; Placebo BID with treatment extension to VDPHL01 QD and Placebo QD

SUMMARY:
This study will evaluate the safety and efficacy of VDPHL01 in male subjects with Androgenetic Alopecia (AGA).

AGA (or male pattern baldness) is a genetic disorder caused by an excessive (too much) hair follicle response to androgens (hormone) that causes hair loss. VDPHL01 8.5 mg Tablet is an investigational oral drug to treat male pattern baldness.

This multi-center, double blind, study will last about 13 months and includes 11 study visits (screening, baseline (day 1), week 2, month 1, month 2, month 4, month 6, month 8, month 10, month 12, month 13).

The first 7 visits will be part of the placebo-controlled period. The next 3 visits will be part of the treatment extension phase. All subjects will receive active drug in the treatment extension phase.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male aged 18-65 years old;
* Subject has a clinical diagnosis of mild to moderate AGA;
* Subject is in good general health and has normal renal and hepatic function;
* Subject is willing to maintain at least 1/4 inch length hair during the study with the same hairstyle, hair length, and hair color throughout the study; maintain consistent use of general hair care products and regimen through the entire study;
* Subject is willing and able to administer the test article as directed read, understand, and complete required questionnaires in English;
* Subject is willing and able to swallow study drug whole;
* Subject agrees to have a micro dot tattoo placed on their scalp;
* Subject agrees to have this area photographed at study visits as indicated in the protocol.

Exclusion Criteria:

* Subject has uncontrolled blood pressure or orthostatic hypotension;
* Subject has symptoms or history of certain heart or thyroid conditions;
* Subject has a history of or active hair loss due to conditions/diseases other than AGA;
* Subject has a current or recent history of dietary or weight changes, including use of GLP-1 agonists;
* Subject has been diagnosed with COVID-19 within 16 weeks of screening;
* Subject has had previous radiation of the scalp;
* Use of any of the following treatments within the indicated washout period before screening:

  * Subject has used hormone replacement therapy or hormonal modulators within 6 months prior to screening
  * Subject has used oral treatments for hair growth or that can affect hair growth, including systemic retinoids, within 6 months of screening
  * Subject has used systemic calcium channel blockers or beta blockers within 12 weeks prior to screening
  * Subject has used systemic cimetidine, ketoconazole, diazoxide, or corticosteroids (including intramuscular, intraarticular, and intralesional injections) within 12 weeks prior to screening
  * Subject has had any scalp procedures, including surgical, laser, light or energy treatments, micro-needling, injections, platelet rich plasma within 6 months prior to screening
  * Subject has used any topical scalp treatments for hair growth within 12 weeks prior to screening
* Subject has used any other therapy with any medication either topical or oral that might, in the investigator's opinion, interfere with the study;
* Subject has any other condition that, in the investigator's opinion, interfere with the study

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 480 (Estimated)
Dates: Start 2024-11-06 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Changes in non-vellus Target Area Hair Counts (TAHC) | Month 6
  Change from baseline in non-vellus TAHC using digital image analysis at Month 6.
Subjects Evaluation of Treatment Benefit | Month 6
  Subjects will rate their treatment benefit by responding to a hair assessment scale. The proportion of subjects by each response category will be reported at Month 6.

CONTACTS AND LOCATIONS:
Overall Officials: Reid Waldman, M.D., Study Chair — Veradermics, Inc.; Timothy Durso, M.D., Study Chair — Veradermics, Inc.
Locations (44):
- United States (44):
  - Site 36, Birmingham, Alabama
  - Site 28, Phoenix, Arizona
  - Site 30, Fort Smith, Arkansas
  - Site 35, Rogers, Arkansas
  - Site 07, Fountain Valley, California
  - Site 02, Fremont, California
  - Site 34, Sherman Oaks, California
  - Site 21, Vista, California
  - Site 05, Castle Rock, Colorado
  - Site 24, Englewood, Colorado
  - Site 17, Aventura, Florida
  - Site 25, Brandon, Florida
  - Site 42, Hollywood, Florida
  - Site 03, Tampa, Florida
  - Site 43, Atlanta, Georgia
  - Site 31, Boise, Idaho
  - Site 23, Rolling Meadows, Illinois
  - Site 15, Indianapolis, Indiana
  - Site 32, New Albany, Indiana
  - Site 27, West Lafayette, Indiana
  - Site 41, Baton Rouge, Louisiana
  - Site 13, Covington, Louisiana
  - Site 12, Metairie, Louisiana
  - Site 22, Brighton, Massachusetts
  - Site 26, Clarkston, Michigan
  - Site 06, New Brighton, Minnesota
  - Site 18, Hackensack, New Jersey
  - Site 37, Kew Gardens, New York
  - Site 38, New York, New York
  - Site 39, Boardman, Ohio
  - Site 11, Columbus, Ohio
  - Site 08, Broomall, Pennsylvania
  - Site 10, Plymouth Meeting, Pennsylvania
  - Site 20, Greensville, South Carolina
  - Site 09, Knoxville, Tennessee
  - Site 16, Murfreesboro, Tennessee
  - Site 04, Nashville, Tennessee
  - Site 40, Bellaire, Texas
  - Site 44, Dallas, Texas
  - Site 14, Houston, Texas
  - Site 19, West Jordan, Utah
  - Site 29, Lynchburg, Virginia
  - Site 33, Seattle, Washington
  - Site 01, Spokane, Washington

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.phlstudy.com/